CLINICAL TRIAL: NCT04019340
Title: The Impact of a Pluridisciplinary Education Program on Venous Leg Ulcer Size Reduction: a Randomized Controlled Trial
Brief Title: The Impact of a Pluridisciplinary Education Program on Venous Leg Ulcer Size Reduction
Acronym: vened
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: School of Health Sciences Geneva (Other)
Responsible Party: Principal Investigator, Sebastian Probst, Professor in tissue viability and wound care, School of Health Sciences Geneva
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: venous leg ulcer education
Record Dates: First submitted 2019-07-10; First posted 2019-07-15 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Patient Empowerment; Venous Leg Ulcer; Interdisciplinary Communication
Keywords: patient education
MeSH Terms: conditions — Patient Participation; Varicose Ulcer | interventions — Educational Status

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Usual care for patients in the CG is defined as visiting the outpatient wound clinic as prescribed by the physician. Wound size measurement, wound care (including dressing and inspection), and questionnaires will be provided by the institute's nurses.
- Education (Other): Usual care as described for the CG will also be provided to the IG (visit to the outpatient wound clinic as prescribed by the physician). Wound size measurement, wound care (including dressing and inspection), and questionnaires will be provided by the institute's nurses. After baseline data collection (T0) and random allocation to the intervention group, this usual care will be enhanced by a pluridisciplinary educational program
  Interventions: Other: Education

INTERVENTIONS:
Other: Education — Usual care as described for the CG will also be provided to the IG. Wound size measurement, wound care, and questionnaires will be provided by the institute's nurses. Usual care will be enhanced by a pluridisciplinary educational program
  Arms: Education

SUMMARY:
Background and rationale: Venous leg ulcers (VLU) are slow healing wounds with a recurrence rate of 70% and a 60% risk of becoming chronic. The estimated VLU prevalence in the general population is 3%. Current therapeutic approaches are multifaceted and focus on reducing wound size and improving wound healing as well as preventing ulcer recurrence. They require a pluridisciplinary team of health care professionals from the domains of nursing, medicine, physiotherapy and nutrition. Approximately 70% of VLU patients have a knowledge deficit in regards to therapeutic measures and have difficulties with adherence to treatment protocols. However, there are no published studies describing and evaluating the impact of pluridisciplinary educational interventions on adherence to the treatment plan and wound size reduction in VLU patients.

Overall objectives: The objectives of the projected study are to evaluate the effectiveness of nurse-led intervention for high-risk patients with VLU in terms of patient knowledge/therapy adherence and to measure the impact of this intervention on wound size reduction and its evolution over time.

Methodology of the planned study: An international multicenter randomized controlled trial with 248 participants in three Swiss French (n= 124) and two Australian (n=124) wound clinics is proposed. The sample size assumptions are based on a two-sided alpha level of 0.05, power of 0.8, and a medium effect size. Univariate and bivariate analysis will be conducted according to the data level and distribution.

Expected results and impact: The findings of this study will generate new knowledge and the results will contribute to VLU clinical practice guidelines to enhance patient adherence to therapy. Our results will not only help improving patients' quality of life, but also contribute to reducing health expenditure.

DETAILED DESCRIPTION:
Background and rationale: Venous leg ulcers (VLU) are slow healing wounds with a recurrence rate of 70% and a 60% risk of becoming chronic. Signs and symptoms such as pain or exudate are not only a burden on those affected but also on the health care system and society in general. The estimated VLU prevalence in the general population is 3%. Treatment cost for VLU is estimated to be 3% of overall health expenditure. Current therapeutic approaches are multifaceted and focus on reducing wound size and improving wound healing as well as preventing ulcer recurrence. Such approaches include compression therapy, leg elevation, specific ankle-exercises and a protein rich diet. They require a pluridisciplinary team of health care professionals from the domains of nursing, medicine, physiotherapy and nutrition. Approximately 70% of VLU patients have a knowledge deficit in regards to therapeutic measures and have difficulties with adherence to treatment protocols. Therefore, it is of utmost importance that the treatment team provides effective patient education and support during the learning phase. However, there are no published studies describing and evaluating the impact of pluridisciplinary educational interventions on adherence to the treatment plan and wound size reduction in VLU patients.

Overall objectives: The objectives of the projected study are to evaluate the effectiveness of nurse-led intervention for high-risk patients with VLU in terms of patient knowledge/therapy adherence and to measure the impact of this intervention on wound size reduction and its evolution over time.

Specific aims: The effectiveness of the intervention will be defined in terms of changes in behavior (altered adherence to compression therapy, elevation therapy, physical activity therapy, ankle exercise therapy, and protein supplement therapy), and in terms of VLU basic awareness acquisition and wound status evaluation. In addition, occurrence of recurrence after healing and incidence of complications (re-hospitalizations) will be measured (frequency and cost).

Methodology of the planned study: An international multicenter randomized controlled trial with 248 participants in three Swiss French (n= 124) and two Australian (n=124) wound clinics is proposed. The study participants will be consecutive patients of the participating clinics who fulfill the inclusion criteria. Wound care will be performed according to the hospital's standard clinical practice guidelines. Allocation to the intervention group (IG) or the control group (CG) will be concealed. The intervention will consist of VLU patient education care bundle giving patients an opportunity to learn about the use of compression bandages, wearing and putting on compression stockings, and will include the importance of physical activity, ankle exercises, leg elevation and a high-protein diet to healing outcomes. An educational brochure summarizing these aspects will be given to the patients of the IG. This group will be supervised by a study nurse, who will not be identical with the nurse in charge of the control group. Due to the intervention being an educational program, the study cannot be blinded either for the participants or the staff performing the intervention. The sample size assumptions are based on a two-sided alpha level of 0.05, power of 0.8, and a medium effect size. Univariate and bivariate analysis will be conducted according to the data level and distribution.

Expected results and impact: The findings of this study will generate new knowledge and the results will contribute to VLU clinical practice guidelines to enhance patient adherence to therapy. Our results will not only help improving patients' quality of life, but also contribute to reducing health expenditure. Additionally, it is in alignment with the National Strategy on the Prevention of Non-Communicable Diseases 2017 - 2024 establishing prevention work for people with enhanced risks and chronic conditions reinforcing protective factors such as diet and exercise. This pluridisciplinary study (engaging experts in nursing, physiotherapy and nutrition) associates two research centers with high-level expertise in the field of wound care that both successfully conducted and published research results.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older,
* an existing diagnosed open VLU,
* ulcer surface >5 cm2 and > 15 cm2,
* proficiency in the French language

Exclusion Criteria:

* Valid informed consent is not or cannot be given

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Wound size reduction | one year
  Measurement of the impact of a pluridisciplinary educative program on the relative Reduction (in %) of wound size in patients with VLU. Wound size will be measured using WoundWorks® imaging device

SECONDARY OUTCOMES:
Self-care | one year
  Self-care score will be evaluated using the validated self care questionnaire (VeLUSET©_FR),
Effective activity | one year
  Effective activity will be measured using GeneActiv device
wound evaluation | one year
  Wound will be evaluated in terms of exudative status, smell, infection status and pain felt. The TIME strategy (T = tissue removal; I = infection control; M = moisture balance; E = edge advancement) proposed by the European Wound Management Association will be applied
Adherence to lifestyle | one year
  Adherence to lifestyle prescriptions, including physical activity, leg elevation, ankle exercises, wearing compression stockings, will be evaluated using a short health questionnaire
general nutritional status | one year
  General nutritional status of patients will be measured using the MNA® questionnaire, a validated assessment tool that identifies people malnourished or at risk of malnutrition
protein intake | one year
  Daily protein intake of participants in g/kg of body weight will be estimated using FFQ questionnaire, a validated tool developed to assess mean nutrient intakes in the population

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian E Probst, Prof, Principal Investigator — University of Applied Sciences and Arts Western Switzerland
Locations (3):
- Switzerland (3):
  - Cité Génération Maison de santé, Onex, Canton of Geneva
  - Centre hospitalier universitaire vaudois, Lausanne, Canton of Vaud
  - University Hospital Geneva, Geneva

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Probst S, Allet L, Depeyre J, Colin S, Buehrer Skinner M. A targeted interprofessional educational intervention to address therapeutic adherence of venous leg ulcer persons (TIEIVLU): study protocol for a randomized controlled trial. Trials. 2019 Apr 29;20(1):243. doi: 10.1186/s13063-019-3333-4. PMID 31036037